CLINICAL TRIAL: NCT04503031
Title: Comparison of the Endotracheal Tube Cuff Pressure Between a Taper-guard Cuffed Nasal Endotracheal Tube and a Cylindrical-shaped Cuffed Nasal Endotracheal Tube After Changing in Position of Head
Brief Title: Comparison of Nasal Taper-guard Cuffed and a Nasal Cylindrical Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-11-043-001
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Endotracheal Tube; Cuff Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cylindrical tube group (Active Comparator): The patient in cylindrical tube group (n=26) were intubated with cylindrical shaped endotracheal tube.
  Interventions: Device: cylindrical endotracheal tube
- tapergaurd tube group (Experimental): The patient in taperguard tube group (n=26) was intubated with TaperGuard endotracheal tube.
  Interventions: Device: TaperGuard endotracheal tube

INTERVENTIONS:
Device: TaperGuard endotracheal tube — TaperGuard endotracheal tube is intubated
  Arms: tapergaurd tube group
Device: cylindrical endotracheal tube — endotracheal tube is intubated
  Arms: cylindrical tube group

SUMMARY:
This study was designed to evaluate the effect of change of head position on the cuff pressure of TaperGaurd endotracheal tube , compared to cylindrical endotracheal tube during oral surgery.

DETAILED DESCRIPTION:
The patient in cylindrical group (n=26) were intubated with cylindrical shaped endotracheal tube (Unomedical, Kedah, Malaysia) and the patient in tapergaurd group (n=26) was intubated with TaperGuard endotracheal tube (Covidien, Athlone, Ireland). The group allocations were informed to the attending anesthesiologist prior to anesthesia. Tracheal intubation was performed with size of inner diameter 7.0 mm endotracheal tube for male and 6.5 mm endotracheal tube for female by the same anesthesiologist. The anesthesiologist measured cuff pressure and distance from endotracheal tube tip to carina during study period.This study was designed to evaluate the effect of change of head position on the cuff pressure of TaperGaurd endotracheal tube, compared to cylindrical endotracheal tube during oral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient who were underwent nasal intubation

Exclusion Criteria:

* history of difficult intubation, limited neck movement, respiratory diseases and body mass index more than 35 kg/m2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Cuff pressure | 5 minutes after change of head position
  Cuff pressure is measured with a manometer (Mallinckrodt Medical, Hennef, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Mr, Principal Investigator — kyungook national university hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No